CLINICAL TRIAL: NCT04406909
Title: Rapid-Cycle Re-Implementation of TRAining Facilities in Norway
Acronym: TRAiN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Norwegian Department of Health and Social Affairs (Other Government)
Responsible Party: Principal Investigator, Michael Bretthauer, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REK 143984
Record Dates: First submitted 2020-05-13; First posted 2020-05-29 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): Access to training at membership training facility
  Interventions: Other: Access to training facility
- No training (No Intervention): No access to training at membership training facility

INTERVENTIONS:
Other: Access to training facility — Access to training facility under national regulations for COVID control
  Arms: Training

SUMMARY:
This study tests the randomized re-opening of training facilities in Norway in relation to the COVID-19 pandemic. The investigators will use the recently developed concept of rapid-cycle randomized implementation to assure fast and safe re-introduction of training facilities by randomized testing of access restriction and measure virus exposure and immunity as well as clinical disease during the intervention to enable safe and timely downgrading of COVID-19 restrictions.

Members of training facilities in Norway age 18 to 64 years without COVID-19 related comorbidity will after informed consent be randomised to either access to training or no access in a first 2-week cycle. Testing for COVID-19 and ascertainment of clinical disease will be performed after the first cycle. If there is no clinically meaningful difference between the arms, new cycles may be implemented subsequently, e.g. with less distancing restrictions or wider age groups.

ELIGIBILITY:
Inclusion Criteria:

* all members of participating training facilities age 18 years or older who are not at increased risk for severe COVID-19 disease (see www.fhi.no for criteria) are eligible for participation if they

  * plan to use the training facility regularly during the project period
  * are willing to adhere to training policies during the project
  * accept assessment of project endpoints
  * approve handling of data for the project

Exclusion Criteria:

* COVId-19 related comorbidity
* Age below 18 years or above 64 years

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4000 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-05-19 (Estimated); Study Completion 2022-05-19 (Estimated)

PRIMARY OUTCOMES:
COVID-19 RNA test positivity | At the end of Cycle 1 (cycle length is 14 days)
  Percentage of COVID-19 RNA positive individuals
Hospital admission for COVID-19 | 7 days after the end of Cycle 1 (cycle length is 14 days)
  Percentage of people admitted to hospital for COVID-19

SECONDARY OUTCOMES:
individuals with COVID-19 antibodies | 14 to 20 days after the end of Cycle 1 (cycle length is 14 days)
  Percentage of individuals with COVID-19 antibodies by blood sampling
Percentage of individuals with health care contacts | 7 days and 3 months after the end of Cycle 1 (cycle length is 14 days)
  Percentage of people who had any contacs with primary or secondary health care services
Need of ventilator treatment after hospital admission for COVID-19 | 7 days and 3 months after the end of Cycle 1 (cycle length is 14 days)
  Percentage of people in need of ventilator after hosital admission for COVID-19
ICU admission for COVID-19 | 7 days and 3 months after the end of Cycle 1 (cycle length is 14 days)
  Percentage of people admitted to the ICU for COVID-19
Cause-specific death | 7 days and 3 months after the end of Cycle 1 (cycle length is 14 days)
  Percentage of people who died, with cause of death (including underlying cause of death)
COVID-19 RNA test positivity in employees at training centres | At the end of Cycle 1 (cycle length is 14 days)
  Percentage of COVID-19 RNA positive employees who worked at the training centres during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Løberg, MD PhD, Principal Investigator — University of Oslo; Mette Kalager, MD PhD, Principal Investigator — University of Oslo
Locations (1):
- SATS Training, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Helsingen LM, Loberg M, Refsum E, Gjostein DK, Wieszczy P, Olsvik O, Juul FE, Barua I, Jodal HC, Herfindal M, Mori Y, Jore S, Lund-Johansen F, Fretheim A, Bretthauer M, Kalager M; TRAiN study group. Covid-19 transmission in fitness centers in Norway - a randomized trial. BMC Public Health. 2021 Nov 16;21(1):2103. doi: 10.1186/s12889-021-12073-0. PMID 34789188